CLINICAL TRIAL: NCT01974050
Title: PregText: Assessing the Feasibility of Monitoring Influenza Vaccine Safety in Pregnant Women Using Text Messaging
Brief Title: PregText: Feasibility of Monitoring Influenza Vaccine Safety in Pregnant Women Using Text Messaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Melissa Stockwell, Assistant Professor of Pediatrics and Population and Family Health, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: AAAM4906
Record Dates: First submitted 2013-10-28; First posted 2013-11-01 (Estimated); Results first posted 2018-02-09 (Actual); Last update posted 2018-03-12 (Actual); Status verified 2018-02

CONDITIONS: Pregnancy
Keywords: Influenza vaccination
MeSH Terms: conditions — Influenza, Human

ARMS (1):
- Text message monitoring (Other): Use of text messaging to monitor post-vaccination
  Interventions: Behavioral: Text message surveillance

INTERVENTIONS:
Behavioral: Text message surveillance

SUMMARY:
In this study, the investigators will prospectively assess fever rates and other adverse events in pregnant women after administration of inactivated influenza vaccine (IIV) using text messaging. The investigators hypothesize that women <20 weeks gestational age who receive IIV will be willing to enroll in a text messaging-based vaccine adverse event monitoring program and will use it to report fever in the post-vaccination period as well as continue to text pregnancy-related outcomes through the end of their pregnancy.

ELIGIBILITY:
Inclusion Criteria:

1. Are pregnant with a gestational age of <20 weeks either by last menstrual period (LMP) and/or ultrasound
2. Are at least 18 years of age
3. Have a visit at a study site during the enrollment period
4. Receive IIV at that visit
5. Have a cell phone with text messaging capabilities
6. Are English or Spanish-speaking
7. Are willing to report via text message through end of pregnancy

Exclusion Criteria:

1. Decision to not continue with pregnancy
2. Any contraindication to receipt of inactivated influenza vaccines
3. Receipt LAIV (live attenuated influenza vaccine) at that visit
4. Previous receipt of IIV in this pregnancy
5. Presence of fever >=100.4F at time of vaccination;
6. Administration of any antipyretic in the 6-hour period prior to vaccination,
7. Stated intent, at time of vaccination, to use prophylactic antipyretics before the development of a fever;
8. Patient only speaks a language other than English or Spanish
9. Patient does not have a cell phone with text messaging
10. Patient's inability to read text messages

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2013-11; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Stockwell, MD MPH, Principal Investigator — Columbia University; Philip LaRussa, MD, Principal Investigator — Columbia University; Maria Cano, MD MPH, Principal Investigator — Centers for Disease Control and Prevention
Locations (1):
- Columbia University, New York, New York, United States

REFERENCES:
- [Result] Stockwell MS, Cano M, Jakob K, Broder KR, Gyamfi-Bannerman C, Castano PM, Lewis P, Barrett A, Museru OI, Castellanos O, LaRussa PS. Feasibility of Text Message Influenza Vaccine Safety Monitoring During Pregnancy. Am J Prev Med. 2017 Sep;53(3):282-289. doi: 10.1016/j.amepre.2017.03.014. Epub 2017 May 8. PMID 28495223
- See also: PubMed link — https://www.ncbi.nlm.nih.gov/pubmed/28495223

RESULTS

PARTICIPANT FLOW:
Groups:
- Text Message Monitoring: Use of text messaging to monitor post-vaccination
  Text message surveillance
Period: Overall Study
Arm/Group | Text Message Monitoring
Started | 166
Completed | 141
Not Completed | 25

BASELINE CHARACTERISTICS:
Arm/Group | Text Message Monitoring
Number analyzed (Participants) | 166
Age, Customized [Count of Participants; unit: Participants]
  19-25 years | 38
  26-34 years | 75
  35-46 years | 53
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 166
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 96
  Not Hispanic or Latino | 70
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 73
  Black | 15
  Asian | 8
  Indigenous Latin American | 7
  Multiracial | 21
  Other | 42

OUTCOME MEASURES:

1. Primary Outcome: Number of Recruited Eligible Pregnant Women <20 Weeks Gestational Age
Description: Number of eligible pregnant women <20 weeks gestational age who receive IIV who will be willing to enroll in a text messaging-based vaccine adverse event monitoring program
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Text Message Monitoring
Number analyzed (Participants) | 207
Participants | 166

2. Secondary Outcome: Number of Participants Who Replied to Text Messaging to Assess Fever Frequency in the d0-2 Post-vaccination With IIV
Description: Number of enrollees who text temperature-related information for the d0-2 period post-vaccination
Time Frame: on vaccination day and the next 2 days (D0-2)
Measure: Number; unit: participants
Arm/Group | Text Message Monitoring
Number analyzed (Participants) | 166
participants | 141

3. Secondary Outcome: Number of Women Enrollees Who Continue to Text Pregnancy-related Outcomes Through the End of Pregnancy
Description: Feasibility of text messaging to monitor pregnancy outcomes through the end of pregnancy: Number of women enrollees who continue to text pregnancy-related outcomes through the end of their pregnancy
Time Frame: 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Text Message Monitoring
Number analyzed (Participants) | 166
Participants | 141

4. Other Pre Specified Outcome: Number of Participants With a Fever in Days 0 to 2 Post-vaccination
Description: Number of participants with any fever on days 0 to 2 post-vaccination
Time Frame: 2 days
Measure: Count of Participants; unit: Participants
Arm/Group | Text Message Monitoring
Number analyzed (Participants) | 166
Participants | 1

5. Other Pre Specified Outcome: Pregnancy Complication
Description: Problems reported during pregnancy
Time Frame: 9 months
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Pregnancy Outcome
Description: Pregnancy outcome including termination, preterm birth, term birth or stillbirth
Time Frame: 9 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Text Message Monitoring
Serious Adverse Events (participants affected / at risk) | 0/166
Other Adverse Events (participants affected / at risk) | 0/166

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes